CLINICAL TRIAL: NCT02954887
Title: A Randomized, Double-blind, Placebo-controlled Trial to Investigate the Efficacy and Safety of Cannabidiol (CBD; GWP42003-P) in Infants With Infantile Spasms Following an Initial Open-label Pilot Study
Brief Title: Phase 3 Trial of Cannabidiol (CBD; GWP42003-P) for Infantile Spasms: Open-label Extension Phase (GWPCARE7)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GWEP15100 Open-label Extension; 2015-004904-50 (EudraCT Number)
Record Dates: First submitted 2016-11-02; First posted 2016-11-04 (Estimated); Results first posted 2020-07-23 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Infantile Spasms
Keywords: GWP42003-P; Cannabidiol
MeSH Terms: conditions — Spasms, Infantile | interventions — Cannabidiol

STUDY DESIGN:
Masking Description: Open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- GWP42003-P (Experimental): Administered orally, up to the target dose recommended by the data safety monitoring committee.
  Participants continue at the target dose, or the highest tolerated dose up to the target dose, for a total of 12 months' treatment.
  Interventions: Drug: GWP42003-P

INTERVENTIONS:
Drug: GWP42003-P — Clear, colorless to yellow solution containing cannabidiol dissolved in the excipients sesame oil and anhydrous ethanol with added sweetener (sucralose) and strawberry flavoring.
  Other Names: CBD; Cannabidiol

SUMMARY:
This trial consists of 3 parts: a pilot safety phase, a pivotal randomized controlled phase, and an open-label extension phase. The open-label extension phase only will be described in this record. All participants will receive GWP42003-P.

ELIGIBILITY:
Only participants who completed the pilot or pivotal phases of the trial may proceed to take part in this open-label extension phase of the trial.

Key eligibility criteria for the blinded phase were as follows:

Key Inclusion Criteria:

* Participant is diagnosed with IS and has failed to respond adequately following treatment with 1 or more approved IS therapies.

Key Exclusion Criteria:

* Participant is currently taking or has taken clobazam or any mammalian target of rapamycin (mTOR) inhibitor within the 2 weeks prior to the screening visit.
* Participant has a QT interval, corrected for heart rate with Bazett's formula (QTcB), of 460 msec or greater on ECG.
* Participant's caregiver is currently giving or has given recreational or medicinal cannabis, or synthetic cannabinoid-based medications, within the 1 month prior to the screening visit.
* Participant's caregiver is unwilling to abstain from giving the participant (including the participant's mother abstaining themselves, if breastfeeding)recreational or medicinal cannabis, or synthetic cannabinoid-based medications (other than the study drug) during the trial.
* Participant has any known or suspected hypersensitivity to cannabinoids or any of the excipients of the study drug, such as sesame oil.
* Participant has significantly impaired hepatic function at the screening visit.
* Participant has received an investigational medicinal product as part of a clinical trial within a minimum of 5 half-lives prior to the screening visit.

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2017-05-12 (Actual); Primary Completion 2019-06-13 (Actual); Study Completion 2019-06-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (5):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - Le Bonheur Children's Hospital, Memphis, Tennessee
  - Valley Health Clinical Research, Winchester, Virginia
- Poland (2):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Centrum Medyczne POMOC, Lodz

RESULTS

PARTICIPANT FLOW:
Groups:
- GWP42003-P OS: Following completion of the Pilot Phase (NCT02953548), participants were eligible to participate in the Open Label Extension Phase. Participants continued on the same dose administered in the Pilot Phase for a maximum of 1 year and completed a 10-day taper after completing the study or withdrawing. Participants were administered GWP42003-P oral solution (OS) orally, twice daily, or three times daily if poorly tolerated. The dosage was split evenly across the two or three daily administrations to equal the target or most tolerable dose.
Period: Overall Study
Arm/Group | GWP42003-P OS
Started | 9
Completed | 2
Not Completed | 7
Not completed — Withdrawal by Subject | 3
Not completed — Lack of Efficacy | 3
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Arm/Group | GWP42003-P OS
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.2 (5.56)
Age, Customized [Count of Participants; unit: Participants]
  Infants and toddlers (28 days-23 months) | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Severe Treatment-emergent Adverse Events (TEAEs)
Description: TEAEs were collected in members of the Safety Population, comprised of all participants who received at least 1 dose of GWP42003-P. TEAEs are defined as all adverse events not present prior to the first investigational medicinal product (IMP) or placebo administration or any event already present that worsened in severity or frequency following IMP.
Time Frame: From signing of informed consent up to Day 417
Population: Safety Analysis Set: all participants who had received ≥ 1 dose of GWP42003-P
Measure: Count of Participants; unit: Participants
Groups:
- GWP42003-P OS: Following completion of the Pilot Phase (NCT02953548), participants were eligible to participate in the Open-label Extension Phase. Participants continued on the same dose administered in the Pilot Phase for a maximum of 1 year and completed a 10-day taper after completing the study or withdrawing. Participants were administered GWP42003-P oral solution (OS) orally, twice daily, or three times daily if poorly tolerated. The dosage was split evenly across the two or three daily administrations to equal the target or most tolerable dose.
Arm/Group | GWP42003-P OS
Number analyzed (Participants) | 9
Participants | 7

2. Primary Outcome: Number of Participants With Any Low or High Hematology Laboratory Parameter Value
Time Frame: Days 19, 29, 43, 71, 127, 211, 295, 379, and 389
Population: Safety Analysis Set. Only participants with evaluable data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P OS
Number analyzed (Participants) | 9
Participants
  Day 19, Low: number analyzed (Participants) | 8
  Day 19, Low | 3
  Day 19, High: number analyzed (Participants) | 8
  Day 19, High | 4
  Day 29, Low: number analyzed (Participants) | 8
  Day 29, Low | 3
  Day 29, High: number analyzed (Participants) | 8
  Day 29, High | 4
  Day 43, Low: number analyzed (Participants) | 6
  Day 43, Low | 1
  Day 43, High: number analyzed (Participants) | 6
  Day 43, High | 2
  Day 71, Low: number analyzed (Participants) | 5
  Day 71, Low | 1
  Day 71, High: number analyzed (Participants) | 5
  Day 71, High | 3
  Day 127, Low: number analyzed (Participants) | 5
  Day 127, Low | 1
  Day 127, High: number analyzed (Participants) | 5
  Day 127, High | 3
  Day 211, Low: number analyzed (Participants) | 3
  Day 211, Low | 1
  Day 211, High: number analyzed (Participants) | 3
  Day 211, High | 2
  Day 295, Low: number analyzed (Participants) | 3
  Day 295, Low | 2
  Day 295, High: number analyzed (Participants) | 3
  Day 295, High | 0
  Day 379, Low: number analyzed (Participants) | 7
  Day 379, Low | 4
  Day 379, High: number analyzed (Participants) | 7
  Day 379, High | 4
  Day 389, Low: number analyzed (Participants) | 6
  Day 389, Low | 1
  Day 389, High: number analyzed (Participants) | 6
  Day 389, High | 4

3. Primary Outcome: Number of Participants With Any Low or High Biochemistry Laboratory Parameter Value
Time Frame: Days 19, 29, 43, 71, 127, 211, 295, 379, and 389
Population: Safety Analysis Set. Only participants with evaluable data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P OS
Number analyzed (Participants) | 9
Participants
  Day 19, Low | 6
  Day 19, High | 7
  Day 29, Low: number analyzed (Participants) | 8
  Day 29, Low | 6
  Day 29, High: number analyzed (Participants) | 8
  Day 29, High | 6
  Day 43, Low: number analyzed (Participants) | 6
  Day 43, Low | 4
  Day 43, High: number analyzed (Participants) | 6
  Day 43, High | 5
  Day 71, Low: number analyzed (Participants) | 5
  Day 71, Low | 2
  Day 71, High: number analyzed (Participants) | 5
  Day 71, High | 4
  Day 127, Low: number analyzed (Participants) | 5
  Day 127, Low | 4
  Day 127, High: number analyzed (Participants) | 5
  Day 127, High | 3
  Day 211, Low: number analyzed (Participants) | 3
  Day 211, Low | 2
  Day 211, High: number analyzed (Participants) | 3
  Day 211, High | 3
  Day 295, Low: number analyzed (Participants) | 3
  Day 295, Low | 2
  Day 295, High: number analyzed (Participants) | 3
  Day 295, High | 3
  Day 379, Low: number analyzed (Participants) | 7
  Day 379, Low | 5
  Day 379, High: number analyzed (Participants) | 7
  Day 379, High | 7
  Day 389, Low: number analyzed (Participants) | 5
  Day 389, Low | 3
  Day 389, High: number analyzed (Participants) | 5
  Day 389, High | 2

4. Primary Outcome: Number of Participants With Any Clinically Relevant Urinalysis Parameter Value
Description: Clinical relevance was determined by the investigator.
Time Frame: Days 19, 29, 43, 71, 127, 211, 295, 379, and 389
Population: Safety Analysis Set. Only participants with evaluable data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P OS
Number analyzed (Participants) | 9
Participants
  Day 19: number analyzed (Participants) | 7
  Day 19 | 0
  Day 29: number analyzed (Participants) | 7
  Day 29 | 0
  Day 43: number analyzed (Participants) | 6
  Day 43 | 0
  Day 71: number analyzed (Participants) | 5
  Day 71 | 1
  Day 127: number analyzed (Participants) | 4
  Day 127 | 0
  Day 211: number analyzed (Participants) | 3
  Day 211 | 0
  Day 295: number analyzed (Participants) | 2
  Day 295 | 0
  Day 379: number analyzed (Participants) | 6
  Day 379 | 0
  Day 389: number analyzed (Participants) | 3
  Day 389 | 0

5. Primary Outcome: Number of Participants With Clinically Significant Electrocardiogram Findings
Description: Clinical significance was determined by the investigator.
Time Frame: From signing of informed consent up to Day 389
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P OS
Number analyzed (Participants) | 9
Participants | 0

6. Primary Outcome: Number of Participants With Clinically Significant Vital Sign Findings
Description: Clinical significance was determined by the investigator.
Time Frame: From signing of informed consent up to Day 389
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P OS
Number analyzed (Participants) | 9
Participants | 0

7. Primary Outcome: Number of Participants With Clinically Significant Physical Examination Findings
Description: Clinical significance was determined by the investigator.
Time Frame: From signing of informed consent up to Day 389
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P OS
Number analyzed (Participants) | 9
Participants | 0

8. Secondary Outcome: Number of Participants Free of Clinical Spasms
Description: Clinical spasms were determined by video-electroencephalography (VEEG) for at least 8 hours and up to 24 hours.
Time Frame: Days 29, 43, 127, 211, 295, and 379
Population: Safety Analysis Set. Only participants with evaluable data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P OS
Number analyzed (Participants) | 9
Participants
  Day 29: number analyzed (Participants) | 8
  Day 29 | 1
  Day 43: number analyzed (Participants) | 6
  Day 43 | 2
  Day 127: number analyzed (Participants) | 4
  Day 127 | 1
  Day 211: number analyzed (Participants) | 3
  Day 211 | 1
  Day 295: number analyzed (Participants) | 2
  Day 295 | 1
  Day 379: number analyzed (Participants) | 7
  Day 379 | 3

9. Secondary Outcome: Percentage of Participants Free of Clinical Spasms
Description: Clinical spasms were determined by VEEG for at least 8 hours and up to 24 hours.
Time Frame: Days 29, 43, 127, 211, 295, and 379
Population: Safety Analysis Set. Only participants with evaluable data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | GWP42003-P OS
Number analyzed (Participants) | 9
percentage of participants
  Day 29: number analyzed (Participants) | 8
  Day 29 | 11.1
  Day 43: number analyzed (Participants) | 6
  Day 43 | 22.2
  Day 127: number analyzed (Participants) | 4
  Day 127 | 11.1
  Day 211: number analyzed (Participants) | 3
  Day 211 | 11.1
  Day 295: number analyzed (Participants) | 2
  Day 295 | 11.1
  Day 379: number analyzed (Participants) | 7
  Day 379 | 33.3

10. Secondary Outcome: Number of Participants With a Resolution of Hypsarrhythmia
Description: Resolution of hypsarrhythmia was determined by VEEG for at least 8 hours and up to 24 hours.
Time Frame: Days 29, 43, 127, 211, 295, and 379
Population: Safety Analysis Set. Only participants with evaluable data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P OS
Number analyzed (Participants) | 9
Participants
  Day 29: number analyzed (Participants) | 8
  Day 29 | 1
  Day 43: number analyzed (Participants) | 6
  Day 43 | 0
  Day 127: number analyzed (Participants) | 4
  Day 127 | 1
  Day 211: number analyzed (Participants) | 3
  Day 211 | 0
  Day 295: number analyzed (Participants) | 2
  Day 295 | 1
  Day 379: number analyzed (Participants) | 7
  Day 379 | 3

11. Secondary Outcome: Percentage of Participants With a Resolution of Hypsarrhythmia
Description: Resolution of hypsarrhythmia was determined by VEEG for at least 8 hours and up to 24 hours.
Time Frame: Days 29, 43, 127, 211, 295, and 379
Population: Safety Analysis Set. Only participants with evaluable data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | GWP42003-P OS
Number analyzed (Participants) | 9
percentage of participants
  Day 29: number analyzed (Participants) | 8
  Day 29 | 11.1
  Day 43: number analyzed (Participants) | 6
  Day 43 | 0
  Day 127: number analyzed (Participants) | 4
  Day 127 | 11.1
  Day 211: number analyzed (Participants) | 3
  Day 211 | 0
  Day 295: number analyzed (Participants) | 2
  Day 295 | 11.1
  Day 379: number analyzed (Participants) | 7
  Day 379 | 33.3

12. Secondary Outcome: Number of Participants Experiencing Spasms and Seizures by Subtype
Description: Caregivers recorded the participant's spasms and seizures by category in a daily diary. Subtypes of spasms and seizure included, clonic, tonic-clonic, myoclonic, focal, and absence.
Time Frame: Days 19, 29, 127, 211, 295, and 379
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P OS
Number analyzed (Participants) | 9
Participants
  Day 19, Clonic | 0
  Day 19, Tonic-Clonic | 0
  Day 19, Atonic | 0
  Day 19, Myoclonic | 0
  Day 19, Focal | 1
  Day 19, Absence | 0
  Day 19, Not Done | 0
  Day 29, Clonic | 0
  Day 29, Tonic-Clonic | 0
  Day 29, Atonic | 0
  Day 29, Myoclonic | 0
  Day 29, Focal | 1
  Day 29, Absence | 0
  Day 29, Not Done | 0
  Day 127, Clonic | 0
  Day 127, Tonic-Clonic | 1
  Day 127, Atonic | 0
  Day 127, Myoclonic | 1
  Day 127, Focal | 0
  Day 127, Absence | 1
  Day 127, No Done | 0
  Day 211, Clonic | 0
  Day 211, Tonic-Clonic | 1
  Day 211, Atonic | 0
  Day 211, Myoclonic | 0
  Day 211, Focal | 0
  Day 211, Absence | 1
  Day 211, Not Done | 0
  Day 295, Clonic | 0
  Day 295, Tonic-Clonic | 1
  Day 295, Atonic | 1
  Day 295, Myoclonic | 0
  Day 295, Focal | 0
  Day 295, Absence | 1
  Day 295, Not Done | 0
  Day 379, Clonic | 1
  Day 379, Tonic-Clonic | 1
  Day 379, Atonic | 0
  Day 379, Myoclonic | 0
  Day 379, Focal | 1
  Day 379, Absence | 1
  Day 379, Not Done | 0

13. Secondary Outcome: Caregiver Global Impression of Change (CGIC)
Description: The CGIC is a single-question assessment completed by the caregiver. The question assessed the status of the participant's condition since treatment start. The caregiver provided a rating on a 7-point scale: 1, very much improved; 2, much Improved; 3, slightly improved; 4, no change; 5, slightly worse; 6, much worse; 7, very much worse.
Time Frame: Baseline; Days 29, 43, 71, 127, 211, 295, and 379
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | GWP42003-P OS
Number analyzed (Participants) | 9
participants
  Day 29, Very Much Improved | 1
  Day 29, Much Improved | 1
  Day 29, Slightly Improved | 5
  Day 29, No Change | 1
  Day 29, Slightly Worse | 0
  Day 29, Much Worse | 0
  Day 29, Very Much Worse | 0
  Day 29, Not Done | 0
  Day 43, Very Much Improved | 2
  Day 43, Much Improved | 1
  Day 43, Slightly Improved | 3
  Day 43, No Change | 0
  Day 43, Slightly Worse | 0
  Day 43, Much Worse | 0
  Day 43, Very Much Worse | 0
  Day 43, Not Done | 0
  Day 71, Very Much Improved | 3
  Day 71, Much Improved | 0
  Day 71, Slightly Improved | 1
  Day 71 No Change | 0
  Day 71, Slightly Worse | 1
  Day 71, Much Worse | 0
  Day 71, Very Much Worse | 0
  Day 71, Not Done | 0
  Day 127, Very Much Improved | 2
  Day 127, Much Improved | 2
  Day 127, Slightly Improved | 0
  Day 127, No Change | 0
  Day 127, Slightly Worse | 0
  Day 127, Much Worse | 0
  Day 127, Very Much Worse | 0
  Day 127, Not Done | 0
  Day 211, Very Much Improved | 1
  Day 211, Much Improved | 2
  Day 211, Slightly Improved | 0
  Day 211, No Change | 0
  Day 211, Slightly Worse | 0
  Day 211, Much Worse | 0
  Day 211, Very Much Worse | 0
  Day 211, Not Done | 0
  Day 295, Very Much Improved | 1
  Day 295, Much Improved | 2
  Day 295, Slightly Improved | 0
  Day 295, No Change | 0
  Day 295, Slightly Worse | 0
  Day 295, Much Worse | 0
  Day 295, Very Much Worse | 0
  Day 295, Not Done | 0
  Day 379, Very Much Improved | 2
  Day 379, Much Improved | 1
  Day 379, Slightly Improved | 3
  Day 379, No Change | 0
  Day 379, Slightly Worse | 1
  Day 379, Much Worse | 1
  Day 379, Very Much Worse | 0
  Day 379, Not Done | 1

14. Secondary Outcome: Physician Global Impression of Change (PGIC)
Description: The PGIC is a single-question assessment completed by the investigator. The question assessed the status of the participant's condition since treatment start. The investigator provided a rating on a 7-point scale: 1, very much improved; 2, much Improved; 3, slightly improved; 4, no change; 5, slightly worse; 6, much worse; 7, very much worse.
Time Frame: Baseline; Days 29, 43, 71, 127, 211, 295, and 379
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | GWP42003-P OS
Number analyzed (Participants) | 9
participants
  Day 29, Very Much Improved | 1
  Day 29, Much Improved | 1
  Day 29, Slightly Improved | 2
  Day 29, No Change | 4
  Day 29, Slightly Worse | 0
  Day 29, Much Worse | 0
  Day 29, Very Much Worse | 0
  Day 29, Not Done | 0
  Day 43, Very Much Improved | 1
  Day 43, Much Improved | 0
  Day 43, Slightly Improved | 4
  Day 43, No Change | 1
  Day 43, Slightly Worse | 0
  Day 43, Much Worse | 0
  Day 43, Very Much Worse | 0
  Day 43, Not Done | 0
  Day 71, Very Much Improved | 1
  Day 71, Much Improved | 2
  Day 71, Slightly Improved | 1
  Day 71, No Change | 1
  Day 71, Slightly Worse | 0
  Day 71, Much Worse | 0
  Day 71, Very Much Worse | 0
  Day 71, Not Done | 0
  Day 127, Very Much Improved | 1
  Day 127, Much Improved | 2
  Day 127, Slightly Improved | 1
  Day 127, No Change | 0
  Day 127, Slightly Worse | 0
  Day 127, Much Worse | 0
  Day 127, Very Much Worse | 0
  Day 127, Not Done | 0
  Day 211, Very Much Improved | 0
  Day 211, Much Improved | 1
  Day 211, Slightly Improved | 1
  Day 211, No Change | 1
  Day 211, Slightly Worse | 0
  Day 211, Much Worse | 0
  Day 211, Very Much Worse | 0
  Day 211, Not Done | 0
  Day 295, Very Much Improved | 0
  Day 295, Much Improved | 1
  Day 295, Slightly Improved | 0
  Day 295, No Change | 1
  Day 295, Slightly Worse | 0
  Day 295, Much Worse | 1
  Day 295, Very Much Worse | 0
  Day 295, Not Done | 0
  Day 379, Very Much Improved | 0
  Day 379, Much Improved | 1
  Day 379, Slightly Improved | 3
  Day 379, No Change | 2
  Day 379, Slightly Worse | 1
  Day 379, Much Worse | 1
  Day 379, Very Much Worse | 0
  Day 379, Not Done | 1

15. Secondary Outcome: Number of Responders
Description: A responder is defined as a participant experiencing a resolution of hypsarrhythmia and free of spasms. Test for responders was conducted by VEEG for at least 8 hours and up to 24 hours.
Time Frame: Days 29, 43, 127, 211, 295, and 379
Population: Safety Analysis Set. Only participants with evaluable data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P OS
Number analyzed (Participants) | 9
Participants
  Day 29: number analyzed (Participants) | 8
  Day 29 | 1
  Day 43: number analyzed (Participants) | 6
  Day 43 | 0
  Day 127: number analyzed (Participants) | 4
  Day 127 | 0
  Day 211: number analyzed (Participants) | 3
  Day 211 | 0
  Day 295: number analyzed (Participants) | 2
  Day 295 | 1
  Day 379: number analyzed (Participants) | 7
  Day 379 | 3

16. Secondary Outcome: Percentage of Responders
Description: as for outcome 15
Time Frame: Days 29, 43, 127, 211, 295, and 379
Population: Safety Analysis Set. Only participants with evaluable data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | GWP42003-P OS
Number analyzed (Participants) | 9
percentage of participants
  Day 29: number analyzed (Participants) | 8
  Day 29 | 11.1
  Day 43: number analyzed (Participants) | 6
  Day 43 | 0
  Day 127: number analyzed (Participants) | 4
  Day 127 | 0
  Day 211: number analyzed (Participants) | 3
  Day 211 | 0
  Day 295: number analyzed (Participants) | 2
  Day 295 | 11.1
  Day 379: number analyzed (Participants) | 7
  Day 379 | 33.3

17. Secondary Outcome: Change From Baseline in Height
Description: A positive change indicates an increase in the average participant's height. A negative change indicates a decrease in the average participant's height. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline (Day 1 of Pilot Study); Days 29, 43, 71, 127, 211, 295, 379, and 389
Population: Safety Analysis Set. Only participants with evaluable data were analyzed.
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | GWP42003-P OS
Number analyzed (Participants) | 9
centimeters
  Baseline (Day 1 of Pilot Study) | 75.04 (9.557)
  Day 29, Open-label Extension (OLE): number analyzed (Participants) | 8
  Day 29, Open-label Extension (OLE) | 0.85 (0.980)
  Day 43, OLE: number analyzed (Participants) | 6
  Day 43, OLE | 0.92 (1.530)
  Day 71, OLE: number analyzed (Participants) | 5
  Day 71, OLE | 3.10 (0.652)
  Day 127, OLE: number analyzed (Participants) | 4
  Day 127, OLE | 3.38 (1.377)
  Day 211, OLE: number analyzed (Participants) | 3
  Day 211, OLE | 5.33 (1.258)
  Day 295, OLE: number analyzed (Participants) | 3
  Day 295, OLE | 8.17 (1.528)
  Day 379, OLE: number analyzed (Participants) | 8
  Day 379, OLE | 5.31 (4.036)
  Day 389, OLE: number analyzed (Participants) | 6
  Day 389, OLE | 3.55 (4.085)

18. Secondary Outcome: Change From Baseline in Body Weight.
Description: A positive change indicates an increase in the average participant's weight. A negative change indicates a decrease in the average participant's weight. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline (Day 1 of Pilot Study); Days 29, 43, 71, 127, 211, 295, 379, and 389
Population: Safety Analysis Set. Only participants with evaluable data were analyzed.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | GWP42003-P OS
Number analyzed (Participants) | 9
kilograms
  Baseline (Day 1 of Pilot Study) | 9.92 (3.245)
  Day 29, OLE: number analyzed (Participants) | 8
  Day 29, OLE | 0.39 (0.309)
  Day 43, OLE: number analyzed (Participants) | 6
  Day 43, OLE | 0.75 (0.809)
  Day 71, OLE: number analyzed (Participants) | 5
  Day 71, OLE | 1.10 (0.430)
  Day 127, OLE: number analyzed (Participants) | 4
  Day 127, OLE | 1.25 (0.420)
  Day 211, OLE: number analyzed (Participants) | 3
  Day 211, OLE | 1.17 (0.503)
  Day 295, OLE: number analyzed (Participants) | 3
  Day 295, OLE | 2.10 (0.889)
  Day 379, OLE | 1.19 (0.862)
  Day 389, OLE: number analyzed (Participants) | 6
  Day 389, OLE | 0.98 (0.637)

19. Secondary Outcome: Change From Baseline in Head Circumference
Description: A positive change indicates an increase in the average participant's head circumference. A negative change indicates a decrease in the average participant's head circumference. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline (Day 1 of PIlot Study); Days 29, 43, 71, 127, 211, 295, 379, and 389
Population: Safety Analysis Set. Only participants with evaluable data were analyzed.
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | GWP42003-P OS
Number analyzed (Participants) | 9
centimeters
  Baseline (Day 1 of Pilot Study) | 44.71 (2.724)
  Day 29, OLE: number analyzed (Participants) | 8
  Day 29, OLE | -0.01 (1.229)
  Day 43, OLE: number analyzed (Participants) | 5
  Day 43, OLE | 0.54 (0.288)
  Day 71, OLE: number analyzed (Participants) | 5
  Day 71, OLE | 0.70 (0.570)
  Day 127, OLE: number analyzed (Participants) | 3
  Day 127, OLE | 1.50 (0.500)
  Day 211, OLE: number analyzed (Participants) | 2
  Day 211, OLE | 0.75 (0.354)
  Day 295, OLE: number analyzed (Participants) | 3
  Day 295, OLE | -0.3 (2.31)
  Day 379, OLE: number analyzed (Participants) | 8
  Day 379, OLE | 1.14 (1.707)
  Day 389, OLE: number analyzed (Participants) | 5
  Day 389, OLE | 0.90 (1.782)

20. Secondary Outcome: Change From Baseline in Vineland Adaptive Behavior Scales, Second Edition (Vineland-II) Score
Description: The Vineland-II scores were assessed by the participant's caregiver. Caregivers were asked to score questions in the following categories: the participant's communication, daily living, physical activity, problem behaviors, and social skills and relationships. Scoring was slightly different for each section, but generally ranged from "usually" (2) to "never" (0). The total score is calculated as the sum of standard scores from the domains and converted into the adaptive behavior composite score (ranging from 20 to 160). Higher scores represent greater levels of functioning, and lower scores represent lower levels of functioning. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline (Day 1 of Pilot Study); Day 211, Day 379
Population: Safety Analysis Set. Only participants with evaluable data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GWP42003-P OS
Number analyzed (Participants) | 9
score on a scale
  Baseline, Day 1 of Pilot Study | 33.6 (37.27)
  Day 211 of OLE: number analyzed (Participants) | 3
  Day 211 of OLE | 6.3 (3.51)
  Day 379 of OLE | -5.4 (23.42)

21. Secondary Outcome: Number of Participants With Relapse of Spasms
Description: Analysis could not be conducted for this outcome measure because the study met No Go Criteria. The Pilot Phase concluded after 9 participants completed treatment and demonstrated continued hypsarrhythmia and spasms on follow-up VEEG. The Pivotal Phase was not initiated; however, participants completing the Pilot Phase could roll into the Open Label Extension Phase for up to 1 year.
Time Frame: Day 16 to Day 379
Population: Safety Analysis Set
Arm/Group | GWP42003-P OS
Number analyzed (Participants) | 0

22. Secondary Outcome: Percentage of Participants With Relapse of Spasms
Description: as for outcome 21
Time Frame: Day 16 to Day 379
Population: Safety Analysis Set
Arm/Group | GWP42003-P OS
Number analyzed (Participants) | 0

23. Secondary Outcome: Average Time to Cessation of Spasms
Description: as for outcome 21
Time Frame: Day 1 to Day 379
Population: Safety Analysis Set
Arm/Group | GWP42003-P OS
Number analyzed (Participants) | 0

24. Secondary Outcome: Average Time to Relapse
Description: as for outcome 21
Time Frame: Day 16 to Day 379
Population: Safety Analysis Set
Arm/Group | GWP42003-P OS
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From signing of informed consent up to Day 417
Description: Treatment-emergent adverse events (TEAEs) were collected in members of the Safety Population, comprised of all participants who received at least 1 dose of GWP42003-P. TEAEs are defined as all adverse events not present prior to the first investigational medicinal product (IMP) or placebo administration or any event already present that worsened in severity or frequency following IMP.
Groups:
- Cannabidiol OS: Following completion of the Pilot Phase (NCT02953548), participants were eligible to participate in the Open Label Extension Phase. Participants continued on the same dose administered in the Pilot Phase for a maximum of 1 year and completed a 10-day taper after completing the study or withdrawing. Participants were administered GWP42003-P oral solution (OS) orally, twice daily, or three times daily if poorly tolerated. The dosage was split evenly across the two or three daily administrations to equal the target or most tolerable dose.
Arm/Group | Cannabidiol OS
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 2/9
Other Adverse Events (participants affected / at risk) | 7/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cannabidiol OS (N=9)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Enterovirus infection (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 2
Rhinovirus infection (Infections and infestations) | 2
Bronchiolitis (Infections and infestations) | 1
Pneumonia bacterial (Infections and infestations) | 1
Pneumonia klebsiella (Infections and infestations) | 1
Urinary tract infection bacterial (Infections and infestations) | 1
Viral upper respiratory infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cannabidiol OS (N=9)
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Pyrexia (General disorders) | 2
Drug tolerance (General disorders) | 1
Irritability (Psychiatric disorders) | 2
Sleep disorder (Psychiatric disorders) | 1
Blood triglycerides increased (Investigations) | 2
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 3
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 2
Somnolence (Nervous system disorders) | 1
Myoclonic epilepsy (Nervous system disorders) | 1
Petit mal epilepsy (Nervous system disorders) | 1
Pupils unequal (Eye disorders) | 1
Deafness (Ear and labyrinth disorders) | 1
Middle ear effusion (Ear and labyrinth disorders) | 1
Gingival pain (Gastrointestinal disorders) | 1
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 1
Scoliosis (Musculoskeletal and connective tissue disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Feeding intolerance (Metabolism and nutrition disorders) | 1
Fluid overload (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Urinary tract infection (Infections and infestations) | 2
Viral infection (Infections and infestations) | 1
Bronchiolitis (Infections and infestations) | 1
Ear infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Viral upper respiratory tract infection (Infections and infestations) | 1

LIMITATIONS AND CAVEATS:
This study met No Go Criteria. The Pilot Phase concluded after 9 participants completed treatment, and the Pivotal Phase was not initiated. Participants completing the Pilot Phase could roll into the Open Label Extension Phase for up to 1 year.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2016-09-20): https://cdn.clinicaltrials.gov/large-docs/87/NCT02954887/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-25): https://cdn.clinicaltrials.gov/large-docs/87/NCT02954887/SAP_001.pdf